CLINICAL TRIAL: NCT01340417
Title: Melatonin Levels in Preterm and Term Newborn Infants
Acronym: MELIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P091108; 2010-A01024-35 (Other: ID-RCB)
Record Dates: First submitted 2011-03-30; First posted 2011-04-22 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2013-09

CONDITIONS: Pregnancy Preterm
Keywords: melatonin; preterm; deficiency; neuroprotection
MeSH Terms: conditions — Premature Birth | interventions — Urination; Blood Specimen Collection; Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one label (Experimental): Measurements of melatonin levels in urine, blood, milk.
  Interventions: Other: Measurements of melatonin levels in urine, blood, milk.

INTERVENTIONS:
Other: Measurements of melatonin levels in urine, blood, milk. — Measurements of melatonin levels in urine, blood, milk.

SUMMARY:
The general goal of the present study is to examine the developmental changes caused by melatonin in preterm and term newborns.

The major brain lesions associated with cerebral palsy and cognitive impairment in preterm infants are periventricular white matter damage (WMD). At the present time, despite major improvements in neonatal care, there are no established therapeutic regimens for the treatment of brain lesions in preterms. Melatonin is secreted by the pineal gland; melatonin's neuroprotective action has been well documented in animal experimental models. Neuroprotection is believed to stem from its direct free radical scavenging, indirect antioxidant activities.

Originality Several reports have described melatonin secretion in older children, but only a few have observed melatonin concentrations during the first year of life. Very little is known about the fetal pineal melatonin synthesis and nothing at what prenatal age melatonin synthesis starts. Premature infants have a 3 months delay in the development of melatonin rhythmicity compared to full-term infants. One study found discordant data with decreasing melatonin value around term. The absence of longitudinal study and the low number of children included make the interpretation difficult of the secretion of melatonin at the newborn.

Hypothesis: Infants born before 28 weeks gestation have melatonin deficiency (50pg/ml), compared to newborns at term (100pg/ml).

Study design: prospective, longitudinal, multicenter trial in 3 Neonatal Intensive Care Units in Ile de France. Specific aim is to compare the developmental changes of melatonin in preterm and term newborns (200 infants and their mothers: 4 groups of 50 infants: 24-27GA +6d ; 28-32 GA +6d ; 33-36 GA +6d ; 37-41 GA +6d). Secondary aims are the following:

* determine Melatonin creatinin excretion in preterm infants
* correlate between serum melatonin secretion and urinary melatonin and 6-sulfatoxymelatonin excretion
* determine endogenous melatonin production in the human pineal
* correlate genetic variations between different levels of melatonin in premature infants
* assess clinical and neurological outcomes at term Clinical impact The present clinical project is part of a translational approach, expected data for infants born before 28 weeks gestation is melatonin deficiency which should participate in determining the potential use of melatonin as a neuroprotectant in human preterm neonates.

DETAILED DESCRIPTION:
The general goal of the present study is to examine the developmental changes caused by melatonin in preterm compared to term newborns. This secretion is studied in child and mother's blood, child's urine, the mother's milk for the women who breastfeed (200 infants and their mothers: 4 groups of 50 infants: 24-27 gestational age (GA) +6d ; 28-32 GA +6d ; 33-36 GA +6d ; 37-41 GA +6d). Secondary aims are the following: determine Melatonin creatinin excretion in preterm infants, correlate between serum melatonin secretion and urinary melatonin and 6-sulfatoxymelatonin excretion, determine endogenous melatonin production in the human pineal, correlate genetic variations between different levels of melatonin in premature infants, assess clinical and neurological outcomes at term.

Study duration for each patient Study duration is one year (inclusion time: 9 months) Duration of mother's inclusion:3 days if delivery between 34 and 41+6d weeks of gestation (two blood samples in maternal vein and umbilical vein after delivery and one mother's milk sample on the third day after delivery, D3) 15 days to 3 months if delivery between 24 and 33+6d weeks of gestation (two blood samples in maternal vein and umbilical vein after delivery and mother's milk sample on the third day after delivery,D10-D15, D30, D60 until term age

Duration of infant's inclusion:

* 3 days if delivery between 34 and 41+6d weeks of gestation (1 blood sample on the third day (D3) after delivery and 4 urinary samples at birth and on D3)
* 15 days to 3 months if delivery between 24 and 33+6d weeks of gestation (blood and urinary samples on the third day after delivery,D10-D15, D30, D60 until term (37-42 weeks gestational age)

Population study All the preterm and term newborns in 3 participating centers, will be evaluated in term of eligibility. Their clinical characteristics will be compared to the criteria of inclusion and exclusion before entering into the study. The inclusion of the preterm from 24 GA is justified by the assumption of responsibility of more in earlier of this population in 2009 (limit of viability from 24 GA and/or birth weight > 500g).

The group of the term infants (37-41 GA +6d) will correspond to the inclusion of new-born babies in good health in maternity.

Descriptive analysis The quantitative variables will be described in the form of average (standard deviation) or median (quartiles) according to their Gaussian nature or not. The qualitative variables will be described by their manpower and frequency.

Analyzes of criteria of judgment The principal analysis will compare the rate of children deprived of melatonin between the 4 groups. This comparison will be carried out by a test of the chi-2 or Fisher if suitable. Nevertheless this analysis will be refined by modeling the plasmatic secretion according to the gestational age and of the hour of melatonin measurement. This modeling will use either a mixed model, or a nonlinear model like the models used into pharmacokinetic. In the same way will be modeled the urinary levels of melatonin and in the mother's milk by taking of account the same parameters as previously and the repetition of the measurements. Some parameters will be used like variables of adjustment like the luminous environment, the preeclampsia, the sex, the intrauterine growth restricted infants, multiple pregnancies, the way of childbirth.

The plan of statistical analysis will be finalized at the end of the study and before data management and will be the subject of Master into biostatistics.

The measurement of cortisol, parameters of the ionogram, urea, creatinin, serotonin will be compared between the 4 groups by using parametric tests (ANOVA) or not parametric (KRUSKALL-Wallis) according to the Gaussian nature or not of the variables. The other measurements (blood, urines) will be described in the course of time according to gestational age.

The analyzes will be carried out with software SAS 9.02 .

Clinical impact:

The present clinical project is part of a translational approach, expected data for infants born before 28 weeks gestation is melatonin deficiency which should participate, in addition with existing data and other ongoing studies in an animal model, in determining the potential use of melatonin as a neuroprotectant in human preterm neonates.

It's important to underline that this study must be considered as an interventional study. Indeed, in this study patients have many takings modality while in common practice patients haven't those takings:

* measurements of melatonin levels in urine, blood, milk
* measurements of Serum Cortisol concentrations and urinary excretion
* measurements of Serum Serotonin level

ELIGIBILITY:
Inclusion Criteria:

* Mother:

  * Consent forms from mother or guardian
  * Age ≥ 18 years
  * Mother Heath insurance
* Newborn:

  * Infants born between 24+0 et 41+6 weeks of gestation
  * Infants with informed consent from mother or guardian and mother's social insurance

Exclusion Criteria:

* Mother:

  * Chronic pathology
  * Treatment: Carbamazepine, betablockers, rifampicin, quinolones, cimetidine, 5-Methoxypsoralen or bergapten, 8- methoxypsoralen (or Methoxsalen), CIRCADIN®
* Newborn :

  * Congenital malformations
  * Dermatosis
  * Treatment: cimetidine

Ages: 24 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 380 (Actual)
Dates: Start 2011-04; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measurements of melatonin levels by radioimmunology | 3 days if delivery between 34 and 41+6d weeks of gestation
  Primary outcomes are measurements of melatonin levels in urine, blood, milk. These procedures will be made by radioimmunology, to limit data variability. The reasoning will be made in coefficient of variation intra-test for a patient.
Measurements of melatonin levels by radioimmunology | 15 days to 3 months if delivery between 24 and 33+6d weeks of gestation
  Primary outcomes are measurements of melatonin levels in urine, blood, milk. These procedures will be made by radioimmunology, to limit data variability. The reasoning will be made in coefficient of variation intra-test for a patient.

SECONDARY OUTCOMES:
Serum Cortisol concentrations and urinary excretion | 3 days if delivery between 34 and 41+6d weeks of gestation
  Serum Cortisol concentrations and urinary excretion
  * Assay will use a volume of 20µl
  * Sensitivity is of 15nmol/l
Serum Cortisol concentrations and urinary excretion | 15 days to 3 months if delivery between 24 and 33+6d weeks of gestation
  Serum Cortisol concentrations and urinary excretion
  * Assay will use a volume of 20µl
  * Sensitivity is of 15nmol/l
Serum Serotonin level | 3 days if delivery between 34 and 41+6d weeks of gestation
  Serum Serotonin level:
  Liquid chromatography methods will be used to measure the serotonin rates (5-hydroxytryptamine, 5 HT) blood. The radioenzymatic techniques of reference will be implemented for the measurement of the enzymatic activities of the way of the melatonin (N-acetyl transferase [NAT or AANAT, EC. 2.3.1.5] and hydroxyindole O-methyltransferase [HIOMT or ASMT, EC. 2.1.1.4]) to the level of the blood plates.
Serum Serotonin level | 15 days to 3 months if delivery between 24 and 33+6d weeks of gestation
  Serum Serotonin level:
  Liquid chromatography methods will be used to measure the serotonin rates (5-hydroxytryptamine, 5 HT) blood. The radioenzymatic techniques of reference will be implemented for the measurement of the enzymatic activities of the way of the melatonin (N-acetyl transferase [NAT or AANAT, EC. 2.3.1.5] and hydroxyindole O-methyltransferase [HIOMT or ASMT, EC. 2.1.1.4]) to the level of the blood plates.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie BIRAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Robert DEBRE, Paris, France

REFERENCES:
- [Result] Biran V, Decobert F, Bednarek N, Boizeau P, Benoist JF, Claustrat B, Barre J, Colella M, Frerot A, Garnotel R, Graesslin O, Haddad B, Launay JM, Schmitz T, Schroedt J, Virlouvet AL, Guilmin-Crepon S, Yacoubi A, Jacqz-Aigrain E, Gressens P, Alberti C, Baud O. Melatonin Levels in Preterm and Term Infants and Their Mothers. Int J Mol Sci. 2019 Apr 27;20(9):2077. doi: 10.3390/ijms20092077. PMID 31035572